CLINICAL TRIAL: NCT02213315
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-dose Study to Evaluate the Pharmacokinetics, Immunogenicity, and Safety of Mavrilimumab in Healthy Japanese Subjects
Brief Title: A Double-blind, Placebo-controlled, Single-dose Study to Evaluate the PK, IM, and Safety in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: D2190C00016
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers, Rheumatoid Arthritis, mavrilimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100mg arm (Experimental): 100mg dose
  Interventions: Drug: 100mg Mavrilimumab
- 150mg arm (Experimental): 150mg dose
  Interventions: Drug: 150mg mavrilimumab
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 100mg Mavrilimumab — 100mg Mavrilimumab
  Arms: 100mg arm
Drug: 150mg mavrilimumab — 150mg mavrilmumab
  Arms: 150mg arm
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A phase 1 randomized, double blind single-dose study to evaluate the PK and immunogenicity of single SC 100 and 150 mg doses of mavrilimumab in healthy adult Japanese subjects.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, parallel group, single-dose study to evaluate the PK, immunogenicity, and safety of mavrilimumab at doses of 100 and 150 mg in healthy adult Japanese subjects. The study will be conducted at one site in Europe and subjects will be randomized in a 5:5:2 ratio to 100, 150mg mavrilimumab and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of Japanese ethnicity
* No evidence of clinically significant respiratory disease

Exclusion Criteria:

* Any condition that, would interfere with the evaluation of the study drug or safety of subjects.
* Subject has a known hypersensitivity to any components of the investigational product.
* History of infection requiring hospitalization or treatment with IV antibiotics within 12 weeks before screening, or evidence of clinically significant active infection.
* Subject has a history or present condition of malignancy.
* Subject has a history or presence of drug addiction (urine test) or has alcohol consumption (breath test) of more than 21 (males) or 14 (females) units of alcohol per week.
* Any blood donation or significant loss of blood within 56 days of study initiation,
* Receipt of live (attenuated) vaccine within the 4 weeks before screening or during the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
PK profile of mavrilimumab | from dosing to day 85
  •Non-compartmental PK parameters following a single-dose of mavrilimumab to analyse •Maximum observed concentration (Cmax); area under the concentration-time curve (AUC); time to maximum concentration (Tmax) and half-life (t1/2) from dosing to Day 85 •The number and percentage of subjects that are ADA positive will be summarized by dose

SECONDARY OUTCOMES:
To evaluate the safety of mavrilimumab | from dosing to day 85
  •The secondary outcome of the study is the safety of mavrilimumab as measured by the frequency and severity of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) from dosing to day 85

CONTACTS AND LOCATIONS:
Overall Officials: malcolm Boyce, BSc MB ChB FRCP FFPM, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Research Site, London, United Kingdom